CLINICAL TRIAL: NCT04613427
Title: Predictors of Rupture Risk of Intracranial Aneurysms - Impact of Lipid Metabolism and Mitochondrial Function
Brief Title: Predictors of Rupture Risk of Intracranial Aneurysms
Acronym: RAPID
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: RAPID
Record Dates: First submitted 2020-09-04; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-09

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Intracranial Aneurysm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unruptured intracranial aneurysm: Patients admitted at Haukeland University Hospital in the study period for treatment of UIA.
- Aneurysmal subarachnoid hemorrhage: Patients admitted at Haukeland University Hospital in the study period for treatment of aSAH.

SUMMARY:
Patients admitted to Haukeland University Hospital with either UIA or aSAH underwent a measurement of bioelectrical impedance and body mass composition using InBody 10. Lipids and lipoproteins were collected from plasma. 60 patients in total were included in the study.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) is a condition mainly caused by the rupture of intracranial aneurysms. The estimated prevalence of intracranial aneurysms in the general population is 1-2%, with an annual incidence of aneurysm rupture causing subarachnoid hemorrhage estimated around 1% in Norway. The mortality rates for aneurysmal subarachnoid hemorrhage (aSAH) are as high as 35%, and for the survivors the condition represents a significant morbidity with long-term cognitive impairment and other challenges. With a mean age of 51-55 years at presentation, the burden, both for the patients themselves and on health care resources, is substantial.

Thus, the risk assessment and management of patients with unruptured intracranial aneurysms (UIA) represents a substantial challenge. The number of patients with incidentally discovered cerebral aneurysms is rapidly growing with the increasing use of non-invasive intracranial magnetic resonance imaging (MRI). Therapy options are endovascular coiling, neurosurgical clipping, or observation. To decide whether to perform a potentially harmful prophylactic procedure or not, better tools to predict the risk of rupture in the given individual are required.

Some risk factors, both for the development of an intracranial aneurysm and for the rupture leading to hemorrhage are identified, such as hypertension, age and smoking. Recent research has shown that obesity and hypercholesterolemia is surprisingly associated with an apparent lower risk of aSAH. However, underlying body composition and dyslipidemic patterns has not yet been explored. Increased knowledge of predictors for aneurysm rupture is required, both to improve the patient care and the decision-making concerning the neurosurgical prevention of aSAH.

In the RAPID project, the investigators aim to identify potential new risk factors for the rupture of intracranial aneurysms by comparing the lipid and lipoprotein profile and the body mass composition in patients with UIA and aSAH.

Direct-segmental multisegmental bioimpedance analysis (DSM-BIA) is a valid tool for the assessment of total body and segmental composition and has shown excellent agreements when compared with dual energy X-ray absorptiometry (DEXA). Body composition will be analysed within day 2 after intervention or surgery using a DSM-BIA scanner (InBody S10, BioSpace Ltd, Seoul, South Korea).

Lipids will be measured enzymatically in ethylenediaminetetraacetic acid (EDTA) plasma/serum on a Hitachi 917 system (Roche Diagnostics GmbH, Mannheim, Germany) using the triacylglycerol (GPO-PAP), cholesterol (CHOD-PAP), HDL-cholesterol plus and LDL-cholesterol plus kit from Roche Diagnostics, and the non-esterifies fatty acid (NEFA FD) kit and the phospholipids kit (Phospholipids FS) from "DiaSys Diagnostic Systems GmbH" (Holzheim, Germany). Glucose will be measured in EDTA-plasma using the Gluco-quant Glucose/HK (GLU) kit from Roche. The total fatty acid composition in EDTA-plasma will be analysed using gas chromatography/mass spectrometry (GC/MS).

Lipoprotein particle size analysis will be performed by proton nuclear magnetic resonance (NMR) spectroscopy. Particle concentrations of lipoproteins of different sizes will be calculated from the measured amplitudes of their spectroscopically lipid methyl group NMR signals. Lipoprotein particle size will be derived from the sum of diameter of each subclass multiplied by its relative mass percentage based on the amplitude of its methyl NMR signal. Particle size analysis will be performed by the Norwegian University of Science and Technology (NTNU).

ELIGIBILITY:
Inclusion Criteria:

* Admitted electively for treatment of unruptured intracranial aneurysm
* Admitted acutely for aneurysmal subarachnoid hemorrhage
* Informed consent form signed by patient or close relative

Exclusion Criteria:

* Pregnant
* Pacemaker
* Subarachnoid hemorrhage without identified aneurysmal rupture
* Unruptured aneurysm with previous SAH/intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Haukeland University Hospital with either aneurysmal subarachnoid hemorrhage or unruptured intracranial aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Anthropometric risk factors of ruptured versus unruptured intracranial aneurysms | The anthropometric data will be collected within 96 hours after admittance, as well as information on the predictors and risk factors from the patient journal.
  The case group with SAH patients will be compared to the control group with UIA patients.
  The anthropometric variables is measured by InBody S10 and includes BMI, waist circumference, visceral fat area, body fat mass, body fat percentage, fat free mass, and skeletal muscle mass. The waist/height ratio will be calculated.
  The data will be analyzed by generalized linear modeling (logistic regression), and the models will be controlled for prognostic factors, including sex, age, hypertension, smoking, alcoholism, statin use, family history of SAH, aneurysm size, diabetes, and cardiovascular disease.

SECONDARY OUTCOMES:
Standard lipid risk factors of ruptured versus unruptured intracranial aneurysms | Blood samples collection within 96 hours after admittance. Calculations will be performed within 3 years after study completion (June 2022).
  The lipid risk factors include levels of triacylglycerols (TAGs), total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C) which will be measured in plasma (mmol/L) non-fasting. From these values, we will calculate the levels of non-HDL-C (TC minus HDL-C) and triacylglycerol-rich lipoprotein cholesterol (TRL-C; non-HDL-C minus LDL-C).
Lipid ratios as risk factors of ruptured versus unruptured intracranial aneurysms | The calculations will be performed prior to statistical analyses within 3 years after study completion (June 2022).
  the ratios TAGs/HDL-C, TC/HDL-C, LDL-C/HDL-C and non-HDL-C/HDL-C will be calculated from measured levels.
Apolipoprotein risk factors of ruptured versus unruptured intracranial aneurysms | Blood samples collection within 96 hours after admittance.
  Apolipoprotein A1 and B levels will be measured in serum non-fasting.
Apolipoprotein A1/B ratio as a risk factor of ruptured versus unruptured intracranial aneurysms | Calculations will be performed within 3 years after study completion (June 2022).
  The ratio Apo-A1/Apo-B will be calculated from measured levels.
Lipoprotein subclass risk factors of ruptured versus unruptured intracranial aneurysms. | Blood samples collection within 96 hours after admittance.
  Particle concentrations (nmol/L) of different lipoprotein subclasses (large, medium-sized and small very low-density lipoprotein (VLDL), intermediate density lipoprotein (IDL), LDL and HDL particles) will be measured in plasma by using proton nuclear magnetic resonance (NMR) spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Christian A Helland, MD PhD, Study Director — Haukeland University Hospital
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lovik K, Laupsa-Borge J, Logallo N, Helland CA. Body composition and rupture risk of intracranial aneurysms. Eur J Med Res. 2024 May 24;29(1):297. doi: 10.1186/s40001-024-01888-3. PMID 38790007